CLINICAL TRIAL: NCT02390687
Title: Evaluation of the Efficacy of Probiotics in Chronic Periodontitis Patients-A Randomized Placebo Controlled Study.
Brief Title: Evaluation of the Efficacy of Probiotics in Chronic Periodontitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Next Gen Pharma India Pvt. Ltd. (Industry)
Collaborators: KVG Medical College and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SUL_PERIO-RG_01
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Placebo Lozenges (3 Lozenges per day; 1 lozenge in morning and 2 lozenges in the night). Each placebo lozenge contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Interventions: Drug: Placebo
- Probiotic Arm (Experimental): L. brevis CD2 Lozenges (3 Lozenges per day; 1 lozenge in morning and 2 lozenges in the night). Each probiotic lozenge contains not less than 1 billion CFU of L. brevis CD2
  Interventions: Drug: Probiotic

INTERVENTIONS:
Drug: Probiotic — Each probiotic lozenge contains not less than 1 billion colony forming unit of Lactobacillus brevis CD2
  Other Names: L. brevis CD2 Lozenges
  Arms: Probiotic Arm
Drug: Placebo — Each placebo lozenge contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Arms: Placebo Arm

SUMMARY:
Periodontitis is an infectious inflammatory disease. Bacteria modulate the inflammatory response and alter the diversity of periodontal disease. In recent years, various host-response modulation therapies have been developed to block the pathways responsible for periodontal tissue breakdown.

There have been significant changes with respect to the effectiveness of, and attitudes towards conventional antimicrobial therapy to combat disease. With the threat of widespread antibiotic resistance rendering many antibiotics useless against important diseases, there is an increased necessity not only to minimise antibiotic use and develop novel non-antibiotic-based treatments, but also to raise the profile of disease prevention. One approach that has gained interest over recent years is the use of probiotic bacteria for oral applications. The rationale for their use in oral health care stems from the increase in evidence that supports their claims for benefit for a range of diseases. Lactobacilli play an important role in the maintenance of health by stimulating the natural immunity as well as by contributing to the balance of the microflora, by interacting with the other members of the flora. The application of health promoting bacteria for therapeutic purposes, is one of the strongest emerging fields. Time has come to shift the paradigm of the treatment from specific bacteria elimination to alteration of the bacterial ecology by using probiotics.

So the purpose of this study is to discover a more promising approach for the treatment of chronic periodontitis .

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed chronic generalized periodontitis
* Need of phase 1 therapy
* Pocket probing depth (PPD) of ≥ 5 mm < 7 mm at two and/or more sites
* Patients with no history of allergies to the drugs to be used

Exclusion Criteria:

* Patients on antibiotics within 3 month prior to study
* Patients with any systemic diseases
* Patients with history of any periodontal therapy within 6 months to trial

Ages: 35 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Periodontal Clinical indices | 8 weeks
  Improvement in periodontal clinical indices, namely, Gingival Index (GI), Bleeding on probing (BOP), Probing Pocket Depth (PPD) and Clinical attachment Loss (CAL).

SECONDARY OUTCOMES:
Change in bone pattern | 8 weeks
  Assessment of changes in bone patterns in bith group using digital radio-graphic technique

CONTACTS AND LOCATIONS:
Overall Officials: Mudnoor M Dayakar, MDS, Principal Investigator — KVG Medical College & Hospital
Locations (1):
- Department of Periodontics, K.V.G. College & Hospital,, Kurunjibhag, Sullia (d.k.), Karnataka, India